CLINICAL TRIAL: NCT00971126
Title: A Phase I/II Study of Sorafenib With Combination of Thalidomide in Advanced or Metastatic Hepatocellular Carcinoma
Brief Title: Study of Sorafenib With Combination of Thalidomide in Hepatocellular Carcinoma (HCC)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Two patients in the first dose level be counted as reaching DLT. DSMB recommend terminated early this trial.
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Cheng-Kung University Hospital (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCOGP-1209
Record Dates: First submitted 2009-07-01; First posted 2009-09-03 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2009-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Group Assignment (Experimental)
  Interventions: Drug: sorafenib (Nexavar®), thalidomide (Thado®)

INTERVENTIONS:
Drug: sorafenib (Nexavar®), thalidomide (Thado®) — Phase I Fixed dose of Sorafenib 800mg/day (400mg, p.o., bid); and Escalation dose of Thalidomide at dose Level I: 50 mg/day (50mg, p.o., qd); Level II: 100 mg/day (50mg, p.o., bid); Level III: 150 mg/day (100mg/50mg, p.o., bid); Level IV: 200 mg/day (100mg, p.o., bid).
  Phase II Fixed dose of Sorafenib 800mg/day (400mg, p.o., bid); and MTD of Thalidomide at phase I study.
  Other Names: Nexavar®), Thado®

SUMMARY:
The purpose of this phase I study is to determine the maximal tolerable dose (MTD) of thalidomide (THADO®) in combination with fixed dose of sorafenib (NEXAVAR®) for the treatment of advanced or metastatic HCC.

The Phase II purpose of this study is to determine the disease control rate (complete response + partial response + stable disease) for at least 4 months of sorafenib (NEXAVAR®) plus phase I determined MTD of thalidomide (THADO®) in patients with advanced or metastatic HCC.

DETAILED DESCRIPTION:
This is a non-randomized, open-labeled, single-arm, multi-center, phase I /II clinical study. The Phase I purpose of this study is to determine the maximal tolerable dose (MTD) of thalidomide (THADO®) in combination with fixed dose of sorafenib (NEXAVAR®) for the treatment of advanced or metastatic HCC, and the dose-limiting toxicity (DLT) profiles and other toxicity profiles in patients receiving fixed dose of sorafenib (NEXAVAR®) plus escalating dose of thalidomide (THADO). The Phase II primary objective of this study is to determine the disease control rate (complete response + partial response + stable disease) for at least 4 months of sorafenib (NEXAVAR®) plus phase I determined MTD of thalidomide (THADO®) in patients with advanced or metastatic HCC. The Phase II secondary objective of this study is to determine the objective tumor response rate, the time to tumor progression, the progression-free survival, the overall survival, and the safety and adverse event profiles, the changes of circulating biomarkers relating to angiogenesis and their correlation with disease control rate.

The sample size are required up to 24 patients for the phase I study and 53 patients for the phase II study.

Sorafenib (NEXAVAR®): supplied to Good Manufacturing Practice standards by Bayer Health Care, Taiwan as a film-coated tablet, each of which contains sorafenib tosylate (274mg) equivalent to 200 mg of sorafenib. Thalidomide (THADO®): supplied to Good Manufacturing Practice standards by TTY Biopharm Co., Ltd. as a white-yellow capsule, each of which contains 50 mg of thalidomide.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age.
* With histologically or cytologically documented HCC or clinically diagnosed HCC.
* Advanced (surgically unresectable and unsuitable for local therapy), and/or metastatic HCC, and/or patient refused local therapy.
* Performance status of ECOG score 0-2.
* Life expectancy of at least 12 weeks.
* At least one tumor lesion that meets both of the following criteria:

  * measurable (must be by CT-scan or MRI) in at least one dimension according to RECIST;
  * the lesion has not been previously treated with local therapy, such as radiation therapy, hepatic arterial (chemo) embolization, radiofrequency ablation, and percutaneous interventional therapy.
* Previous local therapy, such as radiotherapy, hepatic arterial (chemo)embolization, radiofrequency ablation, percutaneous interventional therapy, is allowed but the treatment must be completed at least 4 weeks prior to the baseline scan.
* Patients have adequate bone marrow reserves defined as:

  * ANC ≧ 1,500/μl;
  * Platelets count ≧ 75,000/μl;
  * Hemoglobin ≧ 8.5 g/dl.
* Adequate liver and renal functions defined as:

  * Child-Turcotte-Pugh score of 7 or lower (class A and well-compensated class B);
  * Liver transaminase (ALT) ≦ 5 x upper limit of normal (ULN);
  * Serum total bilirubin ≦ 3mg/dl;
  * Serum albumin ≧ 2.8 g/dl;
  * Prothrombin time (PT)-internal normalized ration (INR) ≦ 2.3 or partial thrombin time (PTT) ≦ 6 seconds above control;
  * Serum creatinine ≦ 1.5 x ULN.
* Women of childbearing potential and men must agree to use adequate contraception, prior to study entry, during treatment, and at least 3 months after last dose of treatment.
* Patients must understand the protocol and sign a written informed consent.

Exclusion Criteria:

* Previous use of systemic anti-cancer therapy for HCC such as chemotherapy, immunotherapy, and targeting therapy within 4 weeks to study entry.
* Patients with prior use of investigational drugs including sorafenib and thalidomide.
* Active cardiac disease, including CHF NYHA class > 2, active CAD, cardiac arrhythmias requiring anti-arrhythmic therapy other than beta-blockers or digoxin, and uncontrolled hypertension.
* Patients with hemorrhagic diathesis or have history of active bleeding with 30 days prior to study entry.
* History of HIV infection.
* Active or uncontrolled infections requiring antibiotics treatment.
* Metastatic brain or leptomeningeal tumours unless the patients is > 6 months from definitive therapy, has negative imaging study within 4 weeks of study entry, and is clinically stable with respect to the tumour at the time of study entry.
* With seizure disorder requiring medication (such as steroids or anti-epileptics).
* History of organ allograft.
* Undergoing renal dialysis.
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bluffer tumours [Ta, Tis & T1] or any cancer curatively treated > 3 years prior to study entry.
* Pregnant or breast-feeding patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-07; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Terms of efficacy assessment: objective tumor response, overall survival, progression-free survival. Terms of safety assessment: adverse effects, laboratory values. | The overall survival will be measured from the time the patient has started protocol treatment to the date of the patient's death. 2. An interim analysis of safety profiles will be reviewed by safety committee.

CONTACTS AND LOCATIONS:
Overall Officials: Chung Hu Chan, MD, PHD, Principal Investigator — National Health Research Institutes, Taiwan
Locations (1):
- Ghang-Gung Memorial Hospital at Chia-Yi, Chiayi City, Taiwan